CLINICAL TRIAL: NCT06253221
Title: A Randomized, Double-blind, Placebo-controlled Clinical Study to Evaluate Mavacamten in Adolescents (Age 12 Years to < 18 Years) With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Brief Title: A Study to Evaluate Mavacamten in Adolescents With Symptomatic Obstructive Hypertrophic Cardiomyopathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV027-010; 2023-505650-17-00 (Other: EU CTR); U1111-1290-1175 (Other: WHO)
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cardiomyopathy, Hypertrophic
Keywords: HCM; mavacamten; Obstructive Hypertrophic Cardiomyopathy; SCOUT; SCOUT-HCM; Pediatric HCM; Pediatric hypertrophic cardiomyopathy; Symptomatic HCM; oHCM
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — MYK-461

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mavacamten (Experimental): Participants assigned to this arm will receive mavacamten (1 mg to 15 mg) from day 1 to end of treatment at week 200.
  Interventions: Drug: Mavacamten
- Placebo (Experimental): Participants assigned to this arm will receive mavacamten (1 mg to 15 mg) from week 28 to end of treatment at week 200.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mavacamten — Specified dose on specified days
  Other Names: BMS-986427
  Arms: Mavacamten
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and pharmacokinetics of mavacamten in adolescent patients with symptomatic obstructive hypertrophic cardiomyopathy (HCM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HCM
* Presence of LVOT obstruction
* Presence of symptoms

Exclusion Criteria:

* Phenocopy diseases resulting in myocardial hypertrophy not related to sarcomere dysfunction
* Evidence of LVEF <50% in prior 6 months
* Planned escalation in HCM therapy or upcoming intervention (eg, major cardiac surgery, HCM medication dose increase)

Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2031-03-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Valsalva left ventricular outflow tract (LVOT) (VLVOT) gradient | At Week 28

SECONDARY OUTCOMES:
Change from baseline in resting LVOT gradient | At Week 28
Change from baseline in post-exercise peak LVOT gradient | At Week 28
Change from baseline in maximal wall thickness | At Week 28
Change from baseline in ratio between early mitral inflow velocity and mitral annular early diastolic velocity (E/e') | At Week 28
Proportion of participants achieving an increase from baseline to Week 28 in peak oxygen uptake test (pVO2) | From baseline up to Week 28
Proportion of participants achieving a reduction from baseline to Week 28 in maximal LVOT gradient to < 30 mmHg | From baseline up to Week 28
Proportion of participants with at least 1 class improvement in New York Heart Association (NYHA) class from baseline to Week 28 | From baseline up to Week 28
Proportion of participants with at least 1 grade improvement in mitral regurgitation at Week 28 | From baseline up to Week 28
Number of participants with treatment-emergent adverse events (TEAEs) | Up to Week 218
Number of participants with treatment-emergent serious adverse events (TESAEs) | Up to Week 218
Change from baseline in electrocardiogram (ECG) (QT interval) | At Week 28
Number of participants with left ventricular ejection fraction (LVEF) ≤ 30% | Up to Week 200
Number of participants with LVEF < 50% | Up to Week 200
Trough observed plasma concentration (Ctrough) | Up to Week 200
Post-dose plasma concentration of mavacamten | Up to Week 200
Maximum observed concentration (Cmax) | Up to Week 200
Area under the concentration-time curve (AUC) | Up to Week 200
Proportion of participants who evaluate taste and swallowability as neutral or better using taste and swallowability scales | At Day 1 and Week 11
Change from baseline in the Hypertrophic Cardiomyopathy Symptom Questionnaire - Shortness of Breath (HCMSQ SoB) domain | At Week 28

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (47):
- United States (31):
  - Local Institution - 0017, Birmingham, Alabama
  - Local Institution - 0050, Phoenix, Arizona
  - Local Institution - 0032, Los Angeles, California
  - Local Institution - 0008, Los Angeles, California
  - Local Institution - 0033, Palo Alto, California
  - Local Institution - 0044, San Diego, California
  - Local Institution - 0038, Aurora, Colorado
  - Local Institution - 0031, St. Petersburg, Florida
  - Local Institution - 0053, Atlanta, Georgia
  - Local Institution - 0013, Chicago, Illinois
  - Local Institution - 0009, Indianapolis, Indiana
  - Local Institution - 0043, Boston, Massachusetts
  - Local Institution - 0002, Ann Arbor, Michigan
  - Local Institution - 0037, St Louis, Missouri
  - Local Institution - 0052, Morristown, New Jersey
  - Local Institution - 0010, New Hyde Park, New York
  - Local Institution - 0024, New York, New York
  - Local Institution - 0036, New York, New York
  - Local Institution - 0040, The Bronx, New York
  - Local Institution - 0015, Charlotte, North Carolina
  - Local Institution - 0039, Durham, North Carolina
  - Local Institution - 0019, Cincinnati, Ohio
  - Local Institution - 0001, Cleveland, Ohio
  - Local Institution - 0029, Columbus, Ohio
  - Local Institution - 0030, Philadelphia, Pennsylvania
  - Local Institution - 0005, Pittsburgh, Pennsylvania
  - Local Institution - 0034, Memphis, Tennessee
  - Local Institution - 0045, Austin, Texas
  - Local Institution - 0054, Houston, Texas
  - Local Institution - 0003, Salt Lake City, Utah
  - Local Institution - 0012, Charlottesville, Virginia
- Australia (2):
  - Local Institution - 0020, Sydney, New South Wales
  - Local Institution - 0042, Clayton, Victoria
- Canada (2):
  - Local Institution - 0041, Edmonton, Alberta
  - Local Institution - 0046, Toronto, Ontario
- France (2):
  - Local Institution - 0022, Paris
  - Local Institution - 0026, Pessac
- Germany (2):
  - Local Institution - 0006, Munich, Bavaria
  - Local Institution - 0018, Berlin, State of Berlin
- Local Institution - 0047, Dublin 12, D12 N512, Ireland
- Italy (3):
  - Local Institution - 0016, Florence, FI
  - Local Institution - 0051, Genova, GE
  - Local Institution - 0027, Napoli
- Spain (2):
  - Local Institution - 0014, Barcelona, B
  - Local Institution - 0025, Madrid
- United Kingdom (2):
  - Local Institution - 0049, Belfast, BFS
  - Local Institution - 0007, London

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Rossano J, Canter C, Wolf C, Favatella N, Lockman J, Puli S, Javidialsaadi A, Dyme J, Crevar C, Mital S. Mavacamten in symptomatic adolescent patients with obstructive hypertrophic cardiomyopathy: design of the phase 3 SCOUT-HCM trial. Am Heart J. 2026 Feb;292:107283. doi: 10.1016/j.ahj.2025.107283. Epub 2025 Sep 30. PMID 41038603
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06253221.html